CLINICAL TRIAL: NCT05930327
Title: COIN: A Pilot Study of Cash Transfers to Improve Outcomes in Low-Income Preterm Neonates and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-021011; 852454 (Other: University of Pennsylvania)
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Preterm Birth
Keywords: Preterm Birth; Unconditional Cash Transfers; Parental Stress; Breastfeeding
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Value Cash Transfer (Experimental): Participants in the treatment group will receive four $325 payments. The first payment will be disbursed at the time of enrollment (between birth and 4 weeks of age), and second payment on the infant's one-month birthday, third payment on the infant's two-month birthday, and the fourth payment on the infant's three-month birthdays.
  Interventions: Other: Unconditional Cash Transfer (High-Value)
- Low-Value Cash Transfer (Active Comparator): Participants in the control group will receive four $25 payments. The first payment will be disbursed at the time of enrollment (between birth and 4 weeks of age), and second payment on the infant's one-month birthday, third payment on the infant's two-month birthday, and the fourth payment on the infant's three-month birthdays.
  Interventions: Other: Unconditional Cash Transfer (Low-Value)

INTERVENTIONS:
Other: Unconditional Cash Transfer (High-Value) — Monthly, Unconditional Cash Transfer ($325) for 4-months
  Arms: High-Value Cash Transfer
Other: Unconditional Cash Transfer (Low-Value) — Monthly, Unconditional Cash Transfer ($25) for 4-months
  Arms: Low-Value Cash Transfer

SUMMARY:
The investigators are conducting a pilot randomized controlled trial of unconditional cash transfers among Medicaid-eligible birthing parents of preterm infants in a single neonatal intensive care unit (NICU) in Pennsylvania.

The investigators will measure the feasibility and acceptability of the intervention, birthing parents' lived experiences of having a preterm infant and the impacts of cash transfers, and conduct a preliminary assessment of efficacy on birthing parent psychological stress and ability to invest in their infant's care.

DETAILED DESCRIPTION:
Poverty is an important social determinant of health and contributes to child heath disparities. Among preterm infants, low-income is associated with worse long-term health outcomes. Given the connection between poverty and poor health outcomes, an urgent need exists to move beyond describing health disparities for low-income infants and towards interventions that interrupt these pathways in early childhood to improve outcomes.

A growing body of literature suggests that monthly unconditional cash transfers (UCTs) - no strings attached monthly cash payments - to low-income families may be an effective intervention to reduce poverty and financial stress, improve psychological health, and improve child health outcomes. However, current studies on UCTs focus primarily on term infants or heterogenous samples of children, with only a single pilot delivering direct financial assistance to low-income preterm infants. Thus, despite well-documented disparities in outcomes for low-income preterm infants, the impact of UCTs among low-income preterm infants and their families remains unknown.

Toward that end, the investigators are conducting a pilot randomized controlled trial of unconditional cash transfers among Medicaid-eligible birthing parents of preterm infants in a single NICU in Pennsylvania. The investigators have three specific aims:

Aim 1: To determine the feasibility and acceptability of randomizing high-value ($325/month) and low-value ($25/month) UCTs to low-income birthing parents of preterm infants beginning in the first month of life.

Aim 2: To examine birthing parents' lived experiences managing the financial impact of having a preterm infant and the perceived impact.

Exploratory Aim 3: To conduct a preliminary assessment of the efficacy of monthly UCTs on birthing parent psychological stress and ability to invest in their infant's care, recognizing the pilot is not designed to be powered for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid-insured or uninsured by meets income requirements for Medicaid-eligibility, Over 18 years old, Speaks English or Spanish fluently, Lives in Philadelphia county, Has an infant born >=22 and <36 weeks gestational age

Exclusion Criteria:

* Reports being "highly likely" to move to a different state in the next 12 months, Reports planning to place the infant up for adoption at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Acceptability of randomizing high-value and low-value unconditional cash transfers (UCT) to low income birthing parents of preterm infants. | 1 year
  The investigators define acceptability as greater than or equal to 90% of respondents reporting "agree" to "strongly agree" to each of the 4 measures of acceptability on the follow-up surveys at 2-months.
Feasibility of enrolling caregivers of preterm infants in the study procedures and receipt of UCTs. | 1 year
  The investigators will measure the percentage of eligible subjects enrolled in study procedures, percentage of participants eligible for cash transfers who consented to receive the cash transfers, percentage of participants receiving monthly payments delivered within 1-2 days of the the child's monthly birthday. The investigators define feasibility as greater than 60% of those eligible enrolling in the study procedures, greater than or equal to 90% of those eligible for cash transfers to consent to cash transfers, and greater than or equal to 95% of monthly payments delivered within 1-2 days on either side of the child's monthly birthday. The investigators will additionally measure the attrition rate of survey and follow-up interview completion, aiming for an attrition rate less than or equal to 20%.

SECONDARY OUTCOMES:
Lived experiences of caring for a preterm infant admitted to the neonatal intensive care unit. | 1 year
  Birthing parents' perspectives and measures of birthing parent psychological stress as measured through semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Duncan, MD, Principal Investigator — Children's Hospital of Philadelphia/University of Pennsylvania
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouchelle ZM, Nelin TD, Salazar EG, Ragland S, Uwawuike D, Radack JK, Duncan AF. Unconditional cash transfers to low-income preterm infants and their families: a pilot randomized controlled trial. J Perinatol. 2025 Sep;45(9):1233-1239. doi: 10.1038/s41372-025-02293-2. Epub 2025 Apr 11. PMID 40216998